CLINICAL TRIAL: NCT03871829
Title: A Phase 2 Study of Daratumumab Subcutaneous (Dara-SC) Administration in Combination With Carfilzomib and Dexamethasone (DKd) Compared With Carfilzomib and Dexamethasone (Kd) in Participants With Multiple Myeloma Who Have Been Previously Treated With Daratumumab to Evaluate Daratumumab Retreatment
Brief Title: Daratumumab Retreatment in Participants With Multiple Myeloma Who Have Been Previously Treated With Daratumumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision was made to discontinue the 54767414MMY2065 study as the Data Review Committee recommendation was early stop of the study for futility.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108598; 2018-004185-34 (EudraCT Number); 54767414MMY2065 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-03-11; First posted 2019-03-12 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Carfilzomib+Dexamethasone (Kd) (Active Comparator): Participants will receive carfilzomib 20 milligram per square meter (mg/m^2) intravenously (IV) on Day 1 of Cycle 1 and then 70 mg/m^2 on Days 8 and 15 of Cycle 1 and thereafter on Days 1, 8, 15 of Cycle 2 onwards. Participants will receive dexamethasone 20 mg on Cycle 1 Day 1, a second dose of 20 milligram (mg) will be given on Cycle 1 Day 2 and 40 mg IV or orally on Days 8, 15, 22 for Cycle 1. Patients will then receive dexamethasone 40mg on days 1, 8, 15 and 22 for cycles 2-9, then on Days 1, 8, 15 for Cycle 10 onwards, until death, intolerable toxicity, start of a new treatment for multiple myeloma, withdrawal of consent, or end of the study. The total duration of each cycle is 28 Days.
  Interventions: Drug: Carfilzomib 20 mg/m^2; Drug: Carfilzomib 70 mg/m^2; Drug: Dexamethasone 40 mg; Drug: Dexamethasone 20 mg
- Arm B: Dara-SC in combination with Kd (DKd) (Experimental): Participants will receive daratumumab subcutaneous (Dara-SC) 1800 mg by SC injection on Days 1, 8, 15, 22 for Cycle 1 and 2, Days 1 and 15 for Cycle 3-6, Day 1 for Cycle 7 onwards. Participants will receive carfilzomib 20 mg/m^2 IV on Cycle 1 Day 1 and then 70 mg/m^2 on Day 8 and 15 of Cycle 1 and Days 1, 8 and 15 of Cycle 2. Participants will receive dexamethasone 20 mg on Cycle 1 Day 1, a second dose of 20 milligram (mg) will be given on Cycle 1 Day 2 and 40 mg IV or orally on Days 8, 15, 22 for Cycle 1. Patients will then receive dexamethasone 40mg on days 1, 8, 15 and 22 for cycles 2-9, then on Days 1, 8, 15 for Cycle 10 onwards, until death, intolerable toxicity, start of a new treatment for multiple myeloma, withdrawal of consent, or end of the study. The total duration of each cycle is 28 Days.
  Interventions: Drug: Carfilzomib 20 mg/m^2; Drug: Carfilzomib 70 mg/m^2; Drug: Dexamethasone 40 mg; Drug: Dara-SC 1800 mg; Drug: Dexamethasone 20 mg

INTERVENTIONS:
Drug: Carfilzomib 20 mg/m^2 — Carfilzomib 20 mg/m^2 will be administered intravenously (IV).
Drug: Carfilzomib 70 mg/m^2 — Carfilzomib 70 mg/m^2 will be administered IV.
Drug: Dexamethasone 40 mg — Dexamethasone 40 mg will be administered as IV infusion or orally.
Drug: Dara-SC 1800 mg — Dara-SC 1800 mg will be administered by SC injection.
  Arms: Arm B: Dara-SC in combination with Kd (DKd)
Drug: Dexamethasone 20 mg — Dexamethasone 20 mg will be administered as IV infusion or orally.

SUMMARY:
The purpose of this study is to compare the efficacy (rate of very good partial response [VGPR] or better as best response as defined by the International Myeloma Working Group [IMWG] criteria) of daratumumab subcutaneous (Dara-SC) in combination with carfilzomib and dexamethasone (Kd) with the efficacy of Kd in participants with relapsed refractory multiple myeloma who were previously exposed to daratumumab to evaluate daratumumab retreatment.

DETAILED DESCRIPTION:
For relapsed or refractory multiple myeloma, the treatment is determined on an individual basis. Common standard of care regimens use either a proteasome inhibitor (PI) or an immunomodulatory agent (IMiD) in combination with dexamethasone with or without a monoclonal antibody (mAb) such as daratumumab. After relapse from PIs or IMiDs, patients are often retreated with drugs that have same mechanism of action to which they have been sensitive. The disease becomes refractory and all effective treatment options are exhausted. Daratumumab is a human IgG1 mAb that binds with high affinity to unique epitope on cluster of differentiation 38 (CD38) and attacks tumor cells that overexpress CD38. Study is to determine the efficacy of Dara-SC in combination with carfilzomib and dexamethasone (DKd) in adult participants with relapsed refractory MM who had 1 to 3 prior line(s) of treatment including a line containing daratumumab to evaluate daratumumab retreatment. The MM treatment is determined on an individual basis where patient's age, prior therapy, bone marrow function, co-morbidities, patient preference and time to relapse are considered. Common standard of care regimens use either PI or an IMiD in combination with dexamethasone with or without a mAb. It is a targeted immunotherapy that attacks tumor cells that overexpress CD38, a transmembrane glycoprotein, in a variety of hematological malignancies including multiple myeloma. The study will be conducted in 3 phases: Screening (28 days), Treatment, and Follow-Up. Assessments like chest X-ray, spirometry test, electrocardiogram (ECG), will be performed during Screening phase. During the Treatment Phase, participants will be randomized to receive Kd or DKd. Efficacy assessments like bone marrow examination will be performed. Follow-up will continue until the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a response (partial response or better based on investigator's determination of response by International Myeloma Working Group [IMWG] criteria) to daratumumab-containing therapy with response duration of at least 4 months
* Participants must have progressed from or be refractory to their last line of treatment. Relapsed or refractory disease as defined as: a) Relapsed disease is defined as an initial response to previous treatment, followed by confirmed progressive disease (PD) by IMWG criteria greater than (>) 60 days after cessation of treatment. b) Refractory disease is defined as less than (<) 25 percent (%) reduction in M-protein or confirmed PD by IMWG criteria during previous treatment or >60 days after cessation of treatment
* Received 1 to 3 prior line(s) of treatment of which one contained daratumumab, and completed daratumumab at least 3 months prior to randomization. A single line of therapy may consist of 1 or more agents, and may include induction, hematopoietic stem cell transplantation, and maintenance therapy. Radiotherapy, bisphosphonate, or a single short course of corticosteroids (no more than the equivalent of dexamethasone 40 milligram per day [mg/day] for 4 days) would not be considered prior lines of therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1, or 2
* Women of childbearing potential must have a negative urine or serum pregnancy test at screening within 14 days prior to randomization

Exclusion Criteria:

* Previous treatment with daratumumab within the last 3 months prior to randomization
* Discontinuation of daratumumab due to a daratumumab-related adverse event (AE)
* History of malignancy (other than multiple myeloma) unless all treatment of that malignancy was completed at least 2 years before consent and the patient has no evidence of disease. Further exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or breast, or other non-invasive lesion, that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years
* Allergies, hypersensitivity, or intolerance to daratumumab, hyaluronidase, monoclonal antibodies (mAbs), human proteins, or their excipients, or known sensitivity to mammalian-derived products. Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
* Participant is: a) Known to be seropositive for human immunodeficiency virus (HIV) with one or more of the following: not receiving highly active antiretroviral therapy (ART), had a change in ART within 6 months of the start of screening, receiving ART that may interfere with study treatment, cluster of differentiation (CD)4 count <350 (unit: cells per cubic millimeter of blood) at screening, acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within 6 months of start of screening, and not agreeing to start ART and be on ART >4 weeks plus having HIV viral load <400 copies/milliliters (mL) at end of 4-week period (to ensure ART is tolerated and HIV controlled. b) Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Participants with resolved infection (example: participants who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) levels. Those who are PCR positive will be excluded. c) Known to be seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (108):
- United States (11):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Oncology Institute of Hope and Innovation, Tucson, Arizona
  - American Institute of Research (AIR), Whittier, California
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Karmanos Cancer Institute - Wayne State University, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Baylor Scott and White Health, Dallas, Texas
  - Millennium Oncology, Houston, Texas
- Belgium (2):
  - ZNA Stuivenberg, Antwerp
  - UZ Gent, Ghent
- Brazil (14):
  - Universidade Estadual De Campinas, Campinas
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Universidade Federal de Goias - Hospital das Clinicas da UFG, Goiânia
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Ministerio da Saude Instituto Nacional do Cancer, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - CEHON, Salvador
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Clinica Sao Germano, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Instituto Brasileiro de Controle do Cancer - Sao Camilo Oncologia, São Paulo
- Tom Baker Cancer Centre, Calgary, Alberta, Canada
- Denmark (4):
  - Aarhus University Hospital, Aarhus N
  - Regionshospitalet i Holstebro, Holstebro
  - Haematological Research unit HFE-X OUH., Odense
  - Vejle Hospital, Vejle
- France (14):
  - Hopital Claude Huriez, Lille
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Emile Muller, Mulhouse
  - Hotel Dieu, Nantes
  - Hopitaux Universitaires Est Parisien Hopital Saint Antoine, Paris
  - Hopital de la Pitie Salpetriere, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Fentre F Magendie, Hôpital Haut Leveque, CHU Bordeaux, Pessac
  - Centre Hospitalier Lyon-Sud Service d'hematologie, Pierre-Bénite
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - Chu Rennes Hopital Pontchaillou, Rennes
  - Institut Claudius Regaud, Toulouse
  - CHU Bretonneau, Tours
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (12):
  - Universitaetsklinikum Koelnt, Cologne
  - Universitätsklinik Carl Gustav Carus, Med. Klinik u. Poliklinik I, Dresden
  - Evangelisches Krankenhaus Essen-Werden, Essen
  - Universitatsklinikum Essen, Essen
  - Universitatsklinik Hamburg Eppendorf UKE, Hamburg
  - St. Barbara-Klinik Hamm GmbH, Hamm
  - Praxisklinik für Haematologie und Onkologie Koblenz, Koblenz
  - Universitätsmedizin der Johannes gutenberg-Universität; III. Med. Klinik - Germany, Mainz
  - Onkologische Schwerpunkt Praxis, Saarbrücken
  - Klinikum der Eberhard Karls Universitaet Abt fur innere Med II Haematologie Onkologie Germany, Tübingen
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - Universitätsklinikum Würzburg Med. Klinik U. Poliklinik Ii, Würzburg
- Greece (5):
  - University of Athens - Evaggelismos Hospital (Evangelismos Hospital), Athens
  - Alexandra General Hospital of Athens, Athens Attica
  - University Hospital Of Larissa, Larissa
  - University General Hospital of Rio, Pátrai
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
- Italy (18):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Istituto di Ematologia Seràgnoli azienda ospedaliera univeristaria Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS Azienda Ospedaliera San Martino - IST, Genova
  - San Martino Hospital, Genova
  - Asst Ovest Milanese - Ospedale Di Legnano, Legnano
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale Maggiore della Carita, Novara
  - Casa di Cura La Maddalena, Palermo
  - Ospedale Villa Sofia-Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Universita Degli Studi di Roma Tor Vergata, Roma
  - Sapienza University of Rome, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - ASL ROMA, Roma
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Azienda Ospedaliera Santa Maria, Terni
- Netherlands (2):
  - Albert Schweitzer ziekenhuis-lokatie Dordwijk, Dordrecht
  - Zuyderland Medical Center, Sittard
- Poland (4):
  - Szpital Uniwersytecki nr 2 im. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Szpital Wojewodzki w Opolu, Opole
  - Szpital Magodent, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Russia (7):
  - Emergency Hospital of Dzerzhinsk, Dzerzhinsk
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Ryazan Regional Clinical Hospital, Ryazan
  - Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Oncological dispensary #2, Sochi
  - Oncology Dispensary of Komi Republic, Syktyvkar
- Spain (14):
  - Hosp Clinic de Barcelona, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. de Leon, León
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. de La Paz, Madrid
  - Hosp. Costa Del Sol, Málaga
  - Hosp. Univ. Son Espases, Palma
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. de Canarias, San Cristóbal de La Laguna
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Gral. Univ. de Toledo, Toledo

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Bahlis NJ, Zonder J, Karlin L, Plesner T, Paris L, Wrobel T, Hungria V, Besemer B, Crusoe E, Silkjaer T, Perrot A, Moreau P, Wu KL, Delimpasi S, Dimopoulos MA, Levin MD, Mangiacavalli S, Nnane I, Kim YJ, Krevvata M, Sha L, Wroblewski S, Tuozzo A, Carson R, Facon T. Subcutaneous daratumumab plus carfilzomib and dexamethasone (D-Kd) versus carfilzomib and dexamethasone (Kd) in patients with relapsed/refractory multiple myeloma who received previous daratumumab treatment: LYNX study. Leuk Lymphoma. 2025 Dec;66(14):2685-2696. doi: 10.1080/10428194.2025.2561117. Epub 2025 Oct 3. PMID 41041907

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Carfilzomib+Dexamethasone (Kd): Participants received carfilzomib 20 milligram per meter square (mg/m^2) intravenously (IV) on Cycle 1 Day 1 and then 70 mg/m^2 on Cycle 1 Days 8 and 15, and thereafter on Days 1, 8, 15 from Cycle 2 onwards. Participants received dexamethasone 20 milligrams (mg) on Cycle 1 Days 1 and 2, and 40 mg IV or orally on Days 8, 15, 22 of Cycle 1. Participants then received dexamethasone 40 mg IV or orally on Days 1, 8, 15 and 22 of Cycles 2-9, then on Days 1, 8, 15 from Cycle 10 onwards, until confirmed progressive disease (PD), death, intolerable toxicity, start of a new treatment for multiple myeloma, withdrawal of consent, or end of the study, whichever occurs first. Each cycle of 28 days.
- Arm B: Dara-SC in Combination With Kd (DKd): Participants received daratumumab 1800 mg by SC injection (Dara-SC) on Days 1, 8, 15, 22 of Cycle 1 and 2, Days 1 and 15 of Cycle 3-6, and on Day 1 from Cycle 7 onwards. Participants received carfilzomib 20 mg/m^2 IV on Cycle 1 Day 1 and then 70 mg/m^2 on Cycle 1 Days 8 and 15, and Days 1, 8 and 15 from Cycle 2 onwards. Participants received dexamethasone 20 mg on Cycle 1 Days 1 and 2 and 40 mg IV or orally on Days 8, 15, 22 of Cycle 1. Participants then received dexamethasone 40 mg IV or orally on Days 1, 8, 15 and 22 of Cycles 2-9, then on Days 1, 8, 15 from Cycle 10 onwards, until confirmed PD, death, intolerable toxicity, start of a new treatment for multiple myeloma, withdrawal of consent, or end of the study, whichever occurs first. Each cycle of 28 days.
Period: Overall Study
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
Started | 44 | 44
Treated (Safety Analysis Set) | 43 | 43
Completed | 0 | 0
Not Completed | 44 | 44
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 12 | 8
Not completed — Study terminated by sponsor | 31 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd) | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (8.56) | 66.7 (9.72) | 67 (9.12)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 15 | 16 | 31
  From 65 to 84 years | 26 | 28 | 54
  85 years and over | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 23 | 26 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 5 | 8 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 39 | 36 | 75
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 5 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 1 | 2 | 3
  BRAZIL | 8 | 7 | 15
  CANADA | 0 | 2 | 2
  DENMARK | 0 | 3 | 3
  FRANCE | 2 | 5 | 7
  GERMANY | 0 | 2 | 2
  GREECE | 7 | 5 | 12
  ITALY | 10 | 5 | 15
  NETHERLANDS | 1 | 1 | 2
  POLAND | 2 | 1 | 3
  RUSSIAN FEDERATION | 4 | 6 | 10
  SPAIN | 7 | 4 | 11
  UNITED STATES | 2 | 1 | 3
Refractory status [Count of Participants; unit: Participants] — Population: Here, 'N' (number of subjects analyzed) signifies participants who were evaluable for this baseline characteristics.
  Participants
    Anti-CD38 antibody only: number analyzed (Participants) | 43 | 43 | 86
    Anti-CD38 antibody only | 8 | 7 | 15
    Both PI and IMiD: number analyzed (Participants) | 43 | 43 | 86
    Both PI and IMiD | 10 | 5 | 15
    IMiD + anti-CD38: number analyzed (Participants) | 43 | 43 | 86
    IMiD + anti-CD38 | 11 | 14 | 25
    IMiD only: number analyzed (Participants) | 43 | 43 | 86
    IMiD only | 4 | 1 | 5
    PI + IMiD + anti-CD38: number analyzed (Participants) | 43 | 43 | 86
    PI + IMiD + anti-CD38 | 5 | 4 | 9
    PI only: number analyzed (Participants) | 43 | 43 | 86
    PI only | 0 | 1 | 1
Stage of Disease (ISS) [Count of Participants; unit: Participants] — The International Staging System (ISS) system consists of stage I: beta2-microglobulin less than (<)3.5 milligram per liter (mg/l) and albumin greater than or equal to (>=) 3.5 gram (g) per 100 milliliter (mL) (g/100 mL); stage II: neither stage I nor stage III and stage III: beta2-microglobulin >= 5.5 mg/l. Population: Here, 'N' (number of subjects analyzed) signifies participants who were evaluable for this baseline characteristics.
  Participants
    STAGE I: number analyzed (Participants) | 43 | 44 | 87
    STAGE I | 12 | 24 | 36
    STAGE II: number analyzed (Participants) | 43 | 44 | 87
    STAGE II | 19 | 11 | 30
    STAGE III: number analyzed (Participants) | 43 | 44 | 87
    STAGE III | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Very Good Partial Response (VGPR) or Better Response
Description: Percentage of participants achieving VGPR or better response were reported. VGPR or better rate was defined as the percentage of participants achieving VGPR, complete response (CR), or stringent complete response (sCR) in accordance with the International Myeloma Working Group (IMWG) criteria, during or after the study treatment but before the start of subsequent anti-myeloma therapy. IMWG criteria for VGPR: Serum and urine M-component detectable by immunofixation but not on electrophoresis, or greater than or equal to (>=) 90 percent (%) reduction in serum M-protein plus urine M-protein less than (<) 100 milligram (mg)/24 hours; for CR: Negative immunofixation on the serum and urine, and Disappearance of any soft tissue plasmacytomas (PCs), and <5% PCs in bone marrow; for sCR: CR plus normal free light chain (FLC) ratio, and Absence of clonal PCs by immunohistochemistry, immunofluorescence or 2- to 4- color flow cytometry.
Time Frame: Up to 3 years and 4 months
Population: The response-evaluable analysis set included participants who had confirmed diagnosis of multiple myeloma and measurable disease at baseline or screening visit.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 39 | 41
Percentage of participants | 46.2 (32.3) [32.3 to 60.4] | 48.8 (35.1) [35.1 to 62.6]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieved partial response (PR) or better responses based on the computerized algorithm, in accordance with the IMWG criteria, during or after the study treatment but before the start of subsequent anti-myeloma therapy. IMWG criteria for PR: greater than or equal to (>=)50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or less than (<)200 mg/24 hours; If the serum and urine M-protein were not measurable, a decrease of >=50% in the difference between involved and uninvolved free light chain (FLC) levels was required in place of the M-protein criteria; If serum and urine M-protein were not measurable, and serum free light assay is also not measurable, >=50% reduction in bone marrow plasma cells (PCs) was required in place of M-protein, provided baseline bone marrow plasma cell percentage was >=30%; additionally, if present at baseline, >=50% reduction in the size of soft tissue PCs was also required.
Time Frame: Up to 3 years and 7 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 39 | 41
Percentage of participants | 64.1 (49.7) [49.7 to 76.8] | 75.6 (62.1) [62.1 to 86.1]

3. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Better
Description: Percentage of participants achieving CR or better were reported. CR or better rate was defined as the percentage of participants achieving CR or sCR based on the computerized algorithm, according to IMWG response criteria. IMWG criteria for CR: Negative immunofixation on the serum and urine, and Disappearance of any soft tissue plasmacytomas (PCs), and <5% PCs in bone marrow.
Time Frame: Up to 3 years and 7 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 39 | 41
Percentage of participants | 25.6 [14.6 to 39.6] | 12.2 [4.9 to 23.9]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the duration from the date of randomization to either progressive disease (PD) or death, whichever comes first. IMWG criteria for PD: >=25% from lowest response level in serum M-component (the absolute increase must be >=0.5 gram per deciliter [g/dL]) and/or in urine M-component (the absolute increase must be >=200 mg/24 hour); only in participants without measurable serum and urine M-protein levels: increase of >=25% in the difference between involved and uninvolved free light chain levels and the absolute increase must be >10 mg/dL. BMPC%: the absolute % must be >=10%; definite increase in size of existing bone lesions or soft tissue plasmacytomas; definite development of new bone lesions or soft tissue plasmacytomas; development of hypercalcemia (corrected serum calcium >11.5 milligrams per deciliter (mg/dL) or 2.65 millimoles per liter [mmol/L]) that can be attributed solely to PC proliferative disorder.
Time Frame: Up to 3 years and 7 months
Population: Intent-to-treat (ITT) analysis set included all participants who were randomized in the study. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 27 | 24
months | 10.61 (4.70) [4.70 to 19.88] | 10.74 (7.49) [7.49 to 16.16]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of the participant's death due to any cause.
Time Frame: Up to 3 years and 7 months
Population: ITT analysis set included all participants who were randomized in the study. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 12 | 8
months | NA [25.40 to NA] — Mean and upper limit of 90% CI were not estimable due to insufficient number of events. | NA [27.10 to NA] — Mean and upper limit of 90% CI were not estimable due to insufficient number of events.

6. Secondary Outcome: Percentage of Participants With Negative Minimal Residual Disease (MRD)
Description: Percentage of participants with negative MRD were reported. MRD negativity rate, defined as the percentage of participants who had MRD negative status at 10^-5 by bone marrow aspirate after the date of randomization and prior to PD or subsequent anti-myeloma therapy.
Time Frame: Up to 3 years and 7 months
Population: ITT analysis set included all participants who were randomized in the study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 44 | 44
Percentage of participants | 11.4 (3.8) [3.8 to 24.6] | 6.8 (1.4) [1.4 to 18.7]

7. Secondary Outcome: Time to Next Treatment
Description: Time to next treatment was defined as the time from randomization to the start of the next-line treatment.
Time Frame: Up to 3 years and 7 months
Population: ITT analysis set analysis set included all participants who were randomized in the study. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 21 | 15
months | 20.60 [14.06 to 25.40] | 20.14 [11.33 to NA] — Upper limit of 90% CI were not estimable due to insufficient number of events.

8. Secondary Outcome: Serum Concentrations of Daratumumab
Description: Serum concentrations of daratumumab were assessed. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: Day 1 of Cycles 1, 3, and 7 (each cycle of 28 days) and Follow Up (post treatment Week 8; up to 30.3 months)
Population: Pharmacokinetic (PK) analysis set included all participants who had received at least 1 dose of daratumumab subcutaneous (dara-SC) and had at least 1 post-dose PK sample. Here, 'N' (number of participants analysed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: microgram per milliliters (mcg/mL)
Arm/Group | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 22
microgram per milliliters (mcg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 6
  Cycle 1 Day 1 | 39.1 (44.1)
  Cycle 3 Day 1 | 849 (329)
  Cycle 7 Day 1: number analyzed (Participants) | 19
  Cycle 7 Day 1 | 715 (381)
  Post-treatment Week 8: number analyzed (Participants) | 4
  Post-treatment Week 8 | 85.5 (131)

9. Secondary Outcome: Number of Participants With Anti-recombinant Human Hyaluronidase (rHuPH20) Antibodies
Description: The incidence of anti-rHuPH20 antibodies were summarized for all participants who received at least one dose of Dara-SC and had appropriate plasma samples for detection of antibodies to rHuPH20 (at least 1 sample after the start of the first dose of Dara-SC). This outcome measure was planned to be analyzed for specified arm only.
Time Frame: Up to end of study; up to 30.3 months
Population: The immunogenicity analysis set for dara-SC included all randomized participants who had appropriate samples for detection of the antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 35
Participants | 1

10. Secondary Outcome: Number of Participants With Anti-Daratumumab Antibodies
Description: Number of participants who test positive for anti-daratumumab antibodies were reported. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: Up to end of study; up to 30.3 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B: Dara-SC in Combination With Kd (DKd)
Number analyzed (Participants) | 35
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years and 7 months
Description: Serious and non-serious AEs were analyzed on safety population which included all participants who received at least 1 dose of study treatment; and all-cause mortality was analyzed on IIT set which included all participants who were randomized in the study.
Arm/Group | Arm A: Carfilzomib+Dexamethasone (Kd) | Arm B: Dara-SC in Combination With Kd (DKd)
All-Cause Mortality (participants affected / at risk) | 12/44 | 8/44
Serious Adverse Events (participants affected / at risk) | 20/43 | 12/43
Other Adverse Events (participants affected / at risk) | 39/43 | 37/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Carfilzomib+Dexamethasone (Kd) (N=43) | Arm B: Dara-SC in Combination With Kd (DKd) (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Noninfective sialoadenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 3 (5)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Carfilzomib+Dexamethasone (Kd) (N=43) | Arm B: Dara-SC in Combination With Kd (DKd) (N=43)
Anaemia (Blood and lymphatic system disorders) | 14 (37) | 11 (20)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 4 (5)
Lymphopenia (Blood and lymphatic system disorders) | 8 (14) | 3 (15)
Neutropenia (Blood and lymphatic system disorders) | 4 (6) | 8 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (32) | 16 (77)
Cataract (Eye disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (5) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 4 (8)
Nausea (Gastrointestinal disorders) | 7 (7) | 6 (14)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (9)
Asthenia (General disorders) | 6 (8) | 5 (7)
Catheter site pain (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (4) | 7 (11)
Malaise (General disorders) | 3 (4) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 5 (6)
Pyrexia (General disorders) | 4 (4) | 5 (9)
COVID-19 (Infections and infestations) | 9 (10) | 9 (9)
Nasopharyngitis (Infections and infestations) | 3 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Blood creatinine increased (Investigations) | 2 (2) | 4 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (12) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5)
Headache (Nervous system disorders) | 7 (12) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (4)
Insomnia (Psychiatric disorders) | 6 (11) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (5)
Renal impairment (Renal and urinary disorders) | 5 (5) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 7 (13)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 7 (13) | 11 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03871829/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT03871829/SAP_001.pdf